CLINICAL TRIAL: NCT06001762
Title: The TRADE Study: A Phase 2 Trial to Assess the ToleRability of Abemaciclib Dose Escalation in Patients With Early-Stage HR-positive and HER2-negative Breast Cancer
Brief Title: TRADE: Dose Escalation Tolerability of Abemaciclib in HR+ HER2- Early Stage Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Erica Mayer, MD, MPH, Principle Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-355
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Early-stage Breast Cancer; High Risk Breast Carcinoma
Keywords: Breast Cancer; Early-stage high-risk breast cancer; Early-stage breast cancer; High risk breast carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib; Tamoxifen; Anastrozole; Letrozole; exemestane; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Abemaciclib (Experimental): Study procedures will be conducted as follows:
  * Cycles 1 - 24
    * Days 1 - 28 of 28-day cycle: Predetermined dose of Abemaciclib 2 x per day.
    * Endocrine therapy 1 x per day.
  * In clinic visits with blood tests, questionnaires, and assessments:
    * Day 1 of Cycles 1, 2, and 3
    * Day 15 of Cycles 1 and 2
    * Every three cycles after Cycle 3 Day 1.
  * End of treatment visit with blood tests, questionnaires, assessments, and stool sample collection.
  Interventions: Drug: Abemaciclib; Drug: Tamoxifen; Drug: Anastrozole; Drug: Letrozole; Drug: Exemestane; Drug: LHRH Agonist

INTERVENTIONS:
Drug: Abemaciclib — CDK4 and CDK6 inhibitor, tablet taken orally
Drug: Tamoxifen — Selective estrogen receptor modulator, taken orally per institutional standard of care
Drug: Anastrozole — Non-steroidal aromatase inhibitor, taken orally per institutional standard of care
Drug: Letrozole — Non-steroidal aromatase inhibitor, taken orally per institutional standard of care
Drug: Exemestane — Steroidal aromatase inhibitor, taken orally per institutional standard of care
Drug: LHRH Agonist — Luteinizing hormone-releasing hormone agonist), taken orally per institutional standard of care

SUMMARY:
In this research study, investigators are testing if a dose-increasing strategy for abemaciclib will have less side effects and be better tolerated than the standard dosage of abemaciclib for participants with early-stage high-risk hormone receptor positive breast cancer.

The names of the study drugs involved in this study are:

* Abemaciclib (CDK4 and CDK6 inhibitor)
* Tamoxifen (Selective estrogen receptor modulator)
* Anastrozole/Letrozole (Non-steroidal aromatase inhibitors)
* Exemestane (steroidal aromatase inhibitor)
* LHRH (Gonadotropin-releasing hormone agonist, or Luteinizing hormone-releasing hormone agonist)

DETAILED DESCRIPTION:
This research study is a prospective, single-arm, open label, phase 2 study designed to evaluate if a dose-increasing strategy for abemaciclib will have less side effects and be better tolerated than the standard dosage of abemaciclib for participants with early-stage high-risk hormone receptor positive breast cancer.

This research study involves adjuvant abemaciclib plus endocrine (anti-hormone) therapy that works to target breast cancer. Adjuvant therapy is treatment given after surgery, chemotherapy, and/or radiation therapy.

The U.S. Food and Drug Administration (FDA) has approved abemaciclib as a treatment option for early-stage high-risk hormone receptor breast cancer. The FDA has also approved hormonal therapies as treatment for hormone receptor positive breast cancer.

The research study procedures include screening for eligibility, study treatment including laboratory evaluations and questionnaires, blood tests, tumor biopsies, and stool collections.

Participation in this research study is expected to last for at least 2 years and up to 5 years.

It is expected that about 90 people will take part in this research study.

Eli Lilly and Company is supporting this study by providing funding for the study and supplying the study drug, abemaciclib.

ELIGIBILITY:
Inclusion Criteria:

* Stage II or III node-positive HR+/HER2- breast cancer per local laboratory assessment.
* Eligible participants must be appropriate candidates for adjuvant abemaciclib, per assessment of their treating physician.
* Participants must be candidates for adjuvant endocrine therapy, which may have started before or at time of entry onto the trial. Patient may be receiving adjuvant aromatase inhibitor or tamoxifen, +/- ovarian suppression.
* Participants must have undergone definitive surgery of the primary breast tumor(s) within 16 months of study entry.
* At least 21 days must have elapsed between last dose of chemotherapy and registration. Participants who previously received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≤1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to randomization.
* At least 14 days must have elapsed between end of radiotherapy and day 1 of treatment with abemaciclib. Participants who received prior radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. No radiotherapy should be planned to occur during study therapy.
* At least 14 days must have elapsed since most recent breast surgery prior to registration and patient has recovered from side effects of prior surgery.
* Bilateral or multifocal/multicentric breast cancers that meet eligibility criteria are allowed.
* ECOG performance status 0-1
* Men and women with any menopausal status ≥18 years of age
* Adequate organ function as defined below:

  * Absolute neutrophil count (ANC) ≥ 1500 x 10^9/L
  * Platelets ≥ 100 x 10^9/L
  * Hemoglobin ≥ 8g/dL; patients may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Initial treatment must not begin earlier than the day after the erythrocyte transfusion.
  * Bilirubin ≤ 1.5 x ULN. For patients with Gilbert syndrome, the limit is ≤ 2 x institutional ULN AND direct bilirubin within the normal range of normality.
  * AST/ALT ≤ 3 x institutional ULN
* Premenopausal women must have a negative serum or urine pregnancy test. Pregnancy testing does not need to be pursued in female patients who are:

  * Age > 60 years; or
  * Age < 60 with intact uterus and amenorrhea for 12 consecutive months or more AND FSH/estradiol levels within postmenopausal range; or
  * Status-post bilateral oophorectomy, total hysterectomy, or bilateral tubal ligation.
* Women of child-bearing potential and men with partners of childbearing potential must be willing to employ one highly effective form of nonhormonal contraception (with the exception of hormonal IUDs) or two effective forms of nonhormonal contraception by the patient and/or partner and continue its use for the duration of the study treatment and for 3 months after the last dose of abemaciclib.
* Subject must be able to swallow and retain oral medication.
* Ability to understand and the willingness to sign a written informed consent document.
* Non-English-speaking patients are eligible but will be exempt from patient-completed questionnaires.

Exclusion Criteria:

* Prior treatment with any CDK4/6 inhibitor.
* Patients with node-negative breast cancer are not eligible for the trial.
* Concurrent therapy with other investigational agents.
* Diagnosis of inflammatory breast cancer (T4d).
* History of allergic reactions attributed to abemaciclib or similar chemical or biologic composition or excipients.
* Participants with a history of malignancy are ineligible except in the following circumstances:

  --Individuals with a history of invasive breast cancer are not eligible unless they have been disease-free for a minimum of five years.
* Individuals with a malignancy history other than invasive breast cancer are eligible if they have no active malignancy and are deemed by the investigator to be at low risk for recurrence of that malignancy.
* Individuals with the following cancer history are eligible: adequately treated non- melanoma skin cancers, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS) of the breast, stage 1 grade 1 endometrial carcinoma. Other exceptions may exist following review with the sponsor-investigator
* Serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting uncontrolled Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea) or other conditions that in the opinion of the investigator limit compliance with study requirements.
* History of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
* Any of the following due to teratogenic potential of the study drugs:

  * Pregnant women
  * Nursing women
  * Women of childbearing potential who are unwilling to employ adequate contraception (condoms, diaphragms, IUDS, surgical sterilization, abstinence, etc). Hormonal birth control methods are not permitted.
  * Men who are unwilling to employ adequate contraception (condoms, surgical sterilization, abstinence, etc).
* Receipt of an experimental treatment in a clinical trial within the last 30 days or 5 half-lives, whichever is longer, prior to enrollment, or is currently enrolled in any other type of medical research (for example: medical device) judged by the sponsor-investigator not to be scientifically or medically compatible with this study.
* Active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment) or invasive/ systemic fungal infection\
* For patients with known HIV infection, CD4 baseline count should be evaluated: patients with a CDK count ≥ 350 cells/uL can be enrolled. Participants should be on established anti-retroviral therapy (ART) for at least four weeks and have an HIV viral load less than 400 copies/mL prior to enrollment. Potential pharmacological interactions of the ART with abemaciclib and endocrine therapy must be reviewed, particularly for the effects on CYP3A4.
* Patients with active or chronic Hepatitis B or C are eligible provided they meet liver function laboratory criteria and cannot be on any medication with a known interaction with the study agents.
* Participants receiving any medications or substances that are strong inhibitors or inducers of CYP3A4, including selected herbals (e.g., hypericum) and food (e.g., grapefruit) known for pharmacological interactions, cannot be enrolled, due to interference with the dose-escalation, unless the food or supplement has been discontinued at least after an interval equivalent to 3-5 half-lives of the inhibitor.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Composite Adverse Rate at 3 months | 3 months
  The rate of the composite endpoint will be reported, including disaggregated and combined rates of treatment discontinuations and/or dose reductions at 3 months.

SECONDARY OUTCOMES:
Incidence of Grade 2-4 Diarrhea | Up to 26 weeks
  Incidence of grade 2-4 diarrhea will be reported as frequencies and absolute numbers based on CTCAE5.0.
Composite Rate of Abemaciclib | Up to 25 weeks
  The composite rate will be reported, including disaggregated and combined rates of treatment discontinuations, dose reductions, dose holds, and inability to reach or maintain the target dose.
Incidence of Treatment-Related Adverse Events | Up to 25 weeks
  The incidence of treatment-related adverse events will be reported as frequencies and absolute numbers based on CTCAT5.0.
Rate of Inability to Reach the Full Dose | Up to 25 weeks
  Rate of inability to reach the full dose will be reported as the rate of participants who have never reached the full dose at 150mg BID.
Therapeutic Adherence to Oral Adjuvant Therapy | Up to 25 weeks
  Ratio of the self-reported number of pills taken and number of pills prescribed
Dose Intensity of Abemaciclib | 12 weeks
  Rate of patients at full dose (150mg BID) at 12 w versus those unable to reach full dose

CONTACTS AND LOCATIONS:
Overall Officials: Erica Mayer, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (12):
- United States (12):
  - Stamford Hospital, Stamford, Connecticut
  - Eastern Maine Medical Center (Northern Light), Brewer, Maine
  - New England Cancer Specialists, Scarborough, Maine
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute at Steward St. Elizabeth's, Brighton, Massachusetts
  - Dana-Farber Cancer Institute at Foxborough, Foxborough, Massachusetts
  - Dana-Farber Cancer Institute at Merrimack Valley, Methuen, Massachusetts
  - Dana-Farber Cancer Institute at Milford, Milford, Massachusetts
  - Dana-Farber Cancer Institute at South Shore, South Weymouth, Massachusetts
  - Dana-Farber Cancer Insitute at Londonderry Hospital, Londonderry, New Hampshire

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu